CLINICAL TRIAL: NCT01200316
Title: Rocking Motion: Physiologic Effect on the Surgical Stress Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-0129; NCI-2012-01884 (Registry Identifier: NCI CTRP); 10445215 (Other Grant/Funding Number: NINR)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Gastrointestinal Cancer
Keywords: Colon Cancer; Abdominal Surgery; Stress; Rocking Motion; Salivary Cortisol; Postoperative Ileus
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colonic Neoplasms | interventions — Standard of Care; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (Experimental): Post surgical patient to sit in a non-rocking chair for at least sixty minutes per day, and ambulating at least three times per day.
  Interventions: Procedure: Standard of Care; Behavioral: Questionnaire
- Rocking Motion Group (Experimental): Post surgical patient to rock in a rocking chair in 10-20 minute increments for at least sixty minutes per day, and ambulating at least three times per day.
  Interventions: Procedure: Rocking Chair Motion; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Standard of Care — Post surgical patient to sit in a non-rocking chair for at least sixty minutes per day, and ambulating at least three times per day.
  Arms: Standard of Care Group
Procedure: Rocking Chair Motion — Post surgical patient to rock in a rocking chair in 10-20 minute increments for at least sixty minutes per day, and ambulating at least three times per day.
  Arms: Rocking Motion Group
Behavioral: Questionnaire — Beginning on day of surgery till discharge (3-5 days)
  Other Names: Survey

SUMMARY:
After having abdominal surgery, patients often experience a lack of bowel function that can cause nausea, vomiting, abdominal swelling, pain, and/or discomfort. This is known as "post-operative ileus." Patients are usually not allowed to leave the hospital until their doctor is sure that their bowel function has returned.

The goal of this clinical research study is to compare using a rocking chair to the standard of care in improving post-operative ileus after abdominal surgery.

DETAILED DESCRIPTION:
The standard method used to help the return of bowel function after surgery is to have patient get out of bed, sit in a chair for a period of time, and then begin walking the first day after surgery. Patients are then asked to increase the time they spend sitting in the chair and walking every day. However, it is not clear that this is the best method to assist in the return of normal bowel function. Some studies have shown that rocking in a rocking chair may help normal bowel function to return more quickly.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being assigned to either group:

* If you are in Group A, you will use the "rocking chair method." Beginning the first day after surgery, you will sit in a rocking chair and rock back and forth for 10-20 minutes at a time. This will be done for at least 60 minutes (1 hour) per day, until you pass gas for the first time after surgery. The study staff will show the correct method to rock in the rocking chair and give you time to practice while you are in the clinic.
* If you are in Group B, you will use the standard method only. Beginning the first day after surgery, you will sit in a non-rocking chair for at least 60 minutes each day until you pass gas for the first time after surgery.

No matter what group you are in, you will also be asked to begin walking the first day after surgery until you pass gas for the first time after surgery.

You will wear an activity recorder all day attached to a wrist band in order to record your time spent in bed, in the rocking or non-rocking chair, and an activity monitor around your waist to record the time and distance walked during each 24-hour period. The study staff will show you how to wear this activity recorder. You will be encouraged by the study staff to increase the time spent in the chair and walking each day.

You will be given a pencil and pad of paper to note the date and time you first pass gas after surgery.

Study Tests:

On the day before you have surgery, the following tests and procedures will be performed:

* You will be asked to provide demographic information (such as your age and marital status). This information will be coded to protect your privacy.
* You will complete a questionnaire about any symptoms you may be experiencing. This should take about 10 minutes to complete.
* Saliva will be collected to measure your cortisol level. For this saliva to be collected, you will spit into a tube. The level of cortisol in your saliva is used to measure your response to stress.

Every morning while you are in the hospital and until you pass gas for the first time after surgery:

* You will be asked if you have passed gas.
* Saliva will be collected to measure your cortisol level.
* You will complete the symptom questionnaire.
* It will take about ten minutes to complete the questionnaire and to collect the saliva sample.
* You will perform the exercises described in the "Study Groups" section, depending on which group you are assigned to.

Length of Study:

You will be on study from the first day after surgery until you pass gas (usually about 3-5 days). You will be taken off study if you cannot tolerate rocking in a rocking chair, sitting in a non-rocking chair, or walking, due to discomfort or any other reason.

This is an investigational study. There are no additional costs to you for taking part in this study.

Up to 80 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Speak and read English
3. Scheduled to undergo abdominal surgery
4. Tolerate sitting in a rocking or nonrocking chair
5. Able to ambulate
6. Scheduled to receive epidural or intravenous patient controlled analgesia
7. Cognitively intact
8. Signed a study-specific informed consent prior to study entry
9. May include patients undergoing ileostomy or colostomy reversal

Exclusion Criteria:

1) All others will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of Rocking Chair Motion on Surgical-Induced Stress | 3 - 5 days
  Efficacy of rocking chair motion on surgical-induced stress response as measured by salivary cortisol sample collected each morning in two groups of colon cancer patients recovering from abdominal surgery randomized to receive either a rocking chair motion intervention or standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Xin S. Wang, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org